CLINICAL TRIAL: NCT05820945
Title: Evaluation of a Pharmacist-Led Intervention to Reduce Drug-Related Problems in Patients Included in a Home Healthcare Program: A Pragmatic Randomized Clinical Trial
Brief Title: A Pharmaceutical Intervention to Reduce Drug-Related Problems in a Home Healthcare Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Clara Salom, Clinical Pharmacist, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19/141-P
Record Dates: First submitted 2023-03-21; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Polypharmacy; Potentially Inappropriate Medications
Keywords: Medication reconciliation; Medication review; Pharmacist practice pattern; Primary health care; Domiciliary care; Aged

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups in parallel for the duration of the study: (a) intervention group (medication review), in which the patients will receive pharmacist-led medication review, and change proposals through their physician, and (b) control group, in which the patients will be subjected to usual pharmacotherapy management.
Who Masked: Outcomes Assessor
Masking Description: The intervention will be carried out unblinded for the patients/physicians, and the results will be blindly measured by the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication review group (Experimental): Pharmacist-led medication review at patient level, and change proposals at physician level.
  Interventions: Other: Pharmacist-led medication review
- Control group (No Intervention): Usual pharmacotherapy management.

INTERVENTIONS:
Other: Pharmacist-led medication review — Clinical review by a primary care pharmacist of the primary care clinical history and the pharmacological treatment plan. After the review process, a meeting will be held between the pharmacist and the responsible physician in order to present proposals for pharmacotherapeutic optimization.
  Arms: Medication review group

SUMMARY:
The investigators' hypothesis is that the individualized review of the pharmacotherapeutic plans of patients in a home healthcare program will be effective in improving the quality and safety of treatments. This study aims to evaluate the effectiveness of a standardized pharmaceutical intervention for the review and optimization of pharmacological treatments in ATDOM patients (catalan home healthcare program at primary care level), compared to the usual management.

DETAILED DESCRIPTION:
ATDOM is the catalan home healthcare program at primary care level. Patients in home care program are frequently polymedicated, which entails a high risk of drug-related problems (DRPs). The investigators' hypothesis is that the individualized review of the pharmacotherapeutic plans of ATDOM patients will be effective in improving the quality and safety of treatments, reducing DRPs in terms of indication, adequacy, effectiveness, and safety.

The main objective of this study is therefore to evaluate the effectiveness of a standardized pharmaceutical intervention for the review and optimization of pharmacological treatments in ATDOM patients, compared to the usual management.

Specifically, the investigators want to determine, through a six-month intervention, the effectiveness in reducing DRPs per patient and polypharmacy. Additionally, the investigators will evaluate in the intervention group the implementation of the proposals for change or improvement by the responsible physician.

This is a pragmatic randomized clinical trial with a comparable control group, with prospective follow-up of an intervention for the adequacy of the pharmacological treatment of patients in the ATDOM program assigned to primary care teams of the Camp de Tarragona Primary Care Directorate. PRMs, proposals and implementation will be determined.

A descriptive statistical analysis will be carried out using multivariate adjustments.

If the evaluation results are favorable, widespread implementation of the program would be possible. It could be extended to all ATDOM patients or outpatients in general. Thus, interdisciplinary teamwork would be strengthened to favor the health care continuum.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the home care program
* Sixty-five years of age or older
* Active pharmacological treatment plan with at least one drug

Exclusion Criteria:

* The responsible physician considers that participation may harm the patient

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-09-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Medication-related problems | Baseline and 6 months follow-up
  Change in number of medication-related problems
Medication related-problems per patient | Baseline and 6 months follow-up
  Change in number of medication-related problems per patient
Patients with one or more MRPs | Baseline and 6 months follow-up
  Change in number of patients with one or more MRPs
Drugs per patient | Baseline and 6 months follow-up
  Change in number of concomitant drugs per patient
Polymedicated patients | Baseline and 6 months follow-up
  Change in number of polymedicated patients. We define polypharmacy as the simultaneous use of 8 or more different drugs.

SECONDARY OUTCOMES:
Proposals issued | Baseline
  Number of proposals issued by the pharmacist.
Proposals implemented | 6 months follow-up
  Number of proposals implemented by the physician

CONTACTS AND LOCATIONS:
Overall Officials: Clara Salom Garrigues, Pharm, Principal Investigator — DAP Camp de Tarragona, Institut Català de la Salut.
Locations (1):
- Pharmacy, Camp de Tarragona Health Area, Catalan Health Institute, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying the published results will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of the results in a medical journal.
Access Criteria: The anonymized datasets used and/or analyzed during the current study will be available from the principal investigator on reasonable request.

REFERENCES:
- [Derived] Salom-Garrigues C, Aragones E, Giralt M, Campabadal Prats C, Bejarano-Romero F, Canadell L. Evaluation of a pharmacist-led intervention to reduce drug-related problems in patients included in a home healthcare program: study protocol for a pragmatic randomized clinical trial. BMC Geriatr. 2024 Feb 19;24(1):170. doi: 10.1186/s12877-024-04763-2. PMID 38373937